CLINICAL TRIAL: NCT07218887
Title: A Phase 1/2, Open-Label, Multicenter, Dose Finding and Dose Expansion Study to Investigate the Safety, Tolerability, and Efficacy of ALXN2350 Gene Therapy in Adult Participants With BAG3 Mutation Associated Dilated Cardiomyopathy
Brief Title: ALXN2350 in Adult Participants With BAG3-Associated Dilated Cardiomyopathy
Acronym: DCMRestore
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D7030C00001; 2024-519674-40-00 (Other: EU CT Number)
Record Dates: First submitted 2025-10-17; First posted 2025-10-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: BAG3 Mutation Associated Dilated Cardiomyopathy
Keywords: ALXN2350; Gene Therapy; BAG3 Mutation Associated Dilated Cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ALXN2350 (Experimental): Participants will receive one of three dose levels of ALXN2350 depending on the cohort.
  Interventions: Drug: ALXN2350

INTERVENTIONS:
Drug: ALXN2350 — ALXN2350 is a gene therapy product consisting of an AAV9 capsid containing BAG3 transgene. It is administered as a single intravenous (IV) infusion.

SUMMARY:
This Phase 1/2 study is an open-label, dose finding and dose expansion study investigating the safety, tolerability, and efficacy of a single IV infusion of ALXN2350 in adult participants with BAG3 associated DCM.

ELIGIBILITY:
Inclusion Criteria:

* Pathogenic or likely pathogenic mutation in BAG3
* Medical history of diagnosis of DCM
* Stable combination of HF SoC medications
* Adequate acoustic windows for echocardiography

Exclusion Criteria:

* Presence of antibodies to AAV9
* Presence of a pathogenic or likely pathogenic variant in another gene where that other gene is authoritatively recognized as causal for DCM.
* Decompensated HF

Note: Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2032-01-27 (Estimated); Study Completion 2032-01-27 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Baseline up to Week 78

SECONDARY OUTCOMES:
Part B: Number of Participants With TEAEs and SAEs | Baseline up to Week 78
Parts A and B: Number of Participants With Cardiac Events at Weeks 52 and 78 | Weeks 52 and 78
Parts A and B: Time to the First Event of Death, Heart Transplant, Mechanical Circulating Support, or Aborted Sudden Cardiac Death | Baseline up to Week 78

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Research Site, Birmingham, Alabama
  - Research Site, Boston, Massachusetts
  - Research Site, Portland, Oregon
  - Research Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR